CLINICAL TRIAL: NCT04069286
Title: EFFICACY OF ORAL AROEIRA (Schinus Terebinthifolia Raddi) COMPARED TO OMEPRAZOLE IN PARTICIPANTS DIAGNOSED WITH FUNCTIONAL DYSPEPPSIA: A RANDOMIZED AND DOUBLE-BLIND STUDY
Brief Title: EFFICACY OF ORAL AROEIRA (Schinus Terebinthifolia Raddi) COMPARED TO OMEPRAZOLE IN DYSPEPPSIA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Infan Industria Quimica Farmaceutica Nacional (Industry)
Collaborators: Hospital Universitário Oswaldo Cruz (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HB/F3-001/2019
Record Dates: First submitted 2019-08-20; First posted 2019-08-28 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Dyspepsia
MeSH Terms: conditions — Dyspepsia | interventions — Omeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated Group (Experimental): Active Group with 237 participants undergoing treatment with oral mastic (Schinus terebinthifolia Raddi), 1 tablet of 640 mg + 1 placebo capsule, once a day, for a period of 4 weeks
  Interventions: Drug: Oral Aroeira
- Control Group (Active Comparator): Comparator Group with 237 participants undergoing treatment with omeprazole, 1 20mg capsule + 1 placebo tablet, once a day, for a period of 4 weeks.
  Interventions: Drug: Omeprazole 20Mg Capsule

INTERVENTIONS:
Drug: Oral Aroeira — Active Group oral Aroeira (Schinus terebinthifolia Raddi), 1 tablet of 640 mg + 1 placebo capsule, once a day, for a period of 4 weeks.
  Arms: Treated Group
Drug: Omeprazole 20Mg Capsule — Comparator Group omeprazole, 1 20mg capsule + 1 placebo tablet, once a day, for a period of 4 weeks.
  Arms: Control Group

SUMMARY:
This is a prospective, randomized, double - blind study of 474 male and female volunteers with dyspeppsia diagnosed at the Oswaldo Cruz University Hospital Gastroenterology Outpatient Clinic from March 2025 to March 2027.

Hypothesis:

As a non-inferiority study, the hypothesis is that the use of oral Aroeira (Schinus terebinthifolia Raddi) for the treatment of participants diagnosed with functional dyspepsia efficacy not inferior to therapy based on the use of omeprazole.

DETAILED DESCRIPTION:
This is a prospective, randomized, double - blind study of 474 male and female volunteers with dyspeppsia diagnosed at the Oswaldo Cruz University Hospital Gastroenterology Outpatient Clinic from March 2025 to March 2027.

Hypothesis:

As a non-inferiority study, the hypothesis is that the use of oral Aroeira (Schinus terebinthifolia Raddi) for the treatment of participants diagnosed with functional dyspepsia efficacy not inferior to therapy based on the use of omeprazole.

The initial proposal of the project was a prospective, comparative and double blind study between aroeira and omeprazole together with antibiotic treatment for patients diagnosed with gastritis caused by Helicobacter pylori, whose dosage of aroeira (Schinus terebinthifolia Raddi) was 1 tablet of 640 mg, every 12 hours for 4 weeks and omeprazole was 1 capsule of 20 mg, 12/12h, for 4 weeks.

Due to Anvisa requirements, and taking into account the current rationale for gastritis related to this infection, we analyzed that a project with gastritis without the association with H. pylori would not be ideal. So, we are proposing a comparative study with the same drugs (aroeira versus omeprazole) in evaluating the complete relief of dyspeptic symptoms in Dyspepsia Functional. In this new proposal, the N will be 474 participants, maintaining a 1:1 ratio. Research participants will be those who report at least 1 of the 5 dyspeptic symptoms (nausea, heartburn, pain epigastric pain, abdominal discomfort aggravated/relieved by meals and feeling of early satiety) with onset more than 6 months, lasting at least 3 months and excluding other diagnoses by upper digestive endoscopy (EDA).

Our primary objective will be "Compare the effectiveness of oral mastic (Schinus terebinthifolia Raddi) versus omeprazole in relieving complete description of the symptoms of functional dyspepsia. The secondary objectives will be:

1. Evaluate the improvement in the quality of life of participants with dyspeptic symptoms within each treatment (before and afterwards) and between aroeira versus omeprazole at the end of treatment;
2. Evaluate complaints within each treatment (before and after) and between oral mastic versus omeprazole at the end of the treatment treatment;
3. Evaluate possible adverse events to treatment with oral mastic versus omeprazole therapy reported by the participant.

Clinical Trial Protocol Oral Aroeira medicine (Schinus terebinthifolia Raddi) Version 03 of 14-June-2023 HB-F3-01/2019 Sponsor: INFAN - Indústria Química Farmacêutica Nacional S/A

The dosage of this study will be: 1 tablet of oral Aroeira (Schinus terebinthifolia Raddi) of 640mg, once a day, at least period of 4 weeks, and omeprazole, 1 capsule of 20mg, once a day, for a period of 4 weeks.

ELIGIBILITY:
To be eligible to participate in this study, an individual must meet all of the following criteria:

Report of at least 1 of the 5 dyspeptic symptoms, with onset more than 6 months ago, with at least least 3 months in duration, according to the ROME IV Classification criteria:

* Nausea;
* Heartburn;
* Epigastric pain;
* Abdominal discomfort aggravated/relieved by meals;
* Feeling of early satiety.

Manifestation of the desire to participate in the study in a free and informed manner.

Age range between 18 and 80 years old;

Ability and desire to use an acceptable method of contraception listed below during the study and until the last follow-up visit:

* Women - condoms, oral, topical, injectable or implantable contraceptive medications, Intrauterine Devices (IUDs) with or without hormones and true abstinence that is aligned with the participant's preferred and usual lifestyle (periodic abstinence [e.g., methods of table, ovulation, symptothermic, post-ovulation], declaration of abstinence during the period of study or coitus interruptus are not acceptable methods of true abstinence).
* Women - will be referred to a gynecologist for screening and better definition of the method;
* Men - guidance on condom use.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Complete relief dyspeppsia symptom | 30 days after the first day treatment
  Assessment of the proportion of participants with complete relief of dyspeptic symptoms. Complete relief of symptoms will be considered if the scores obtained in items #3, #5 and #7 of the ROME III questionnaire are lower than or equal to their respective reference values for the diagnosis of each symptom of functional dyspepsia.

SECONDARY OUTCOMES:
Life quality Improvement | 60 days after the first day treatment
  Assessment of the proportion of improvement in quality of life using the SF-36 quality of life questionnaire, taking into account the domains "Functional capacity", "Limitation due to physical aspects", "Pain", "General health status", "Vitality ", "Social aspects", "Emotional aspects" and "Mental health" generating a continuous numerical variable (between 0 and 100, where 0 is bad and 100 is good) corresponding to each domain.

CONTACTS AND LOCATIONS:
Overall Officials: Severino B Santos, PhD, Principal Investigator — Hospital Univeristário Oswaldo Cruz

IPD SHARING:
Plan to Share IPD: No